CLINICAL TRIAL: NCT01727843
Title: Phase III Examining the Topical Application of Tranexamic Acid and Postoperative Blood Loss in Femoral Neck Fractures: a Randomized Control Trial.
Brief Title: Topical Application of Tranexamic Acid and Postoperative Blood Loss in Femoral Neck Fractures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Jeff Yach (Other)
Responsible Party: Sponsor-Investigator, Dr. Jeff Yach, PI, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SURG-263-12; 6007434 (Other: Queen's University REB)
Record Dates: First submitted 2012-11-01; First posted 2012-11-16 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Femoral Neck Fracture
Keywords: fracture; hip; tranexamic acid; topical
MeSH Terms: conditions — Femoral Neck Fractures; Fractures, Bone | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tranexamic acid (Experimental): 3000mg/mL tranexamic acid in saline applied directly to the wound at the end of the surgical procedure.
  Interventions: Drug: Tranexamic Acid
- saline (Placebo Comparator): 3000mg/mL saline applied directly to the wound at the end of the surgical procedure
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Tranexamic Acid — drug and placebo applied topically at end of surgery at hip site.
  Other Names: Cyklokapron
  Arms: tranexamic acid
Other: placebo — applied topically to surgical site in OR.
  Other Names: saline solution
  Arms: saline

SUMMARY:
Tranexamic acid (TA) is a synthetic antifibrinolytic agent. It prevents degradation of fibrin and delays the breakdown of hemostatic clots. It has been demonstrated in multiple studies and meta analyses to decrease blood loss in elective hip and knee arthroplasty. However, concerns about the prothrombotic side effects of systemic administration of TA has hindered the widespread adoption of this medication in orthopaedic patients due to their high risk for thrombotic complications such as deep venous thrombosis and pulmonary embolism Topical application of tranexamic acid has been proposed as a way to mitigate the potential prothrombotic effects of TA. Topical application of TA has been demonstrated to be beneficial in oral and cardiac surgery. Plasma levels of TA have been found to be minimal following topical application, minimizing its potential systemic thromboembolic side effects. TA has been used topically in total knee arthroplasty, with significant reductions in blood loss and no increase in thromboembolic complications8,10. Data on the use of TA in hip fracture surgery is limited, and there are no studies examining topical use of TA in hip fracture surgery.

DETAILED DESCRIPTION:
Our study question is: Does topical tranexamic acid decrease blood loss following hemiarthroplasty of the hip for femoral neck fractures? The type of information collected by the research assistant will consist of estimated blood loss during surgery, length of stay in hospital, any wound infections as well as any thromboembolic side effects (blood clots in legs and/or heart) that may occur. The number of units of red blood cells transfused will be recorded up to and including postoperative day 8. Preoperative hemoglobin and lowest postoperative hemoglobin levels up to and including post-op day 8 will also be collected as well as any use of ambulatory aids will be recorded on presentation to hospital, discharge and 6 weeks post operatively.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture patients
* aged 65 and older.

Exclusion Criteria:

* bilateral femoral neck fracture patient and/or one that is not suited to a hemiarthroplasty repair.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2017-11-03 (Actual); Study Completion 2017-11-03 (Actual)

PRIMARY OUTCOMES:
Blood loss | postop 0-8 days.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Yach, MD, Principal Investigator — Queen's Univeristy
Locations (1):
- Queen's Univeristy, KGH, Kingston, Ontario, Canada